CLINICAL TRIAL: NCT04864743
Title: An Open-Label, Multicenter Evaluation of the Pharmacokinetics，Safety and Tolerability of PEG Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection (FRSW117) in Patients With Severe Hemophilia A.
Brief Title: A Study to Evaluate the Pharmacokinetics，Safety and Tolerability of PEG Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Gensciences lnc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTR20210830
Record Dates: First submitted 2021-04-21; First posted 2021-04-29 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-05

CONDITIONS: Severe Hemophilia A
Keywords: severe Hemophilia A; PEG Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection; Pharmacokinetics; Efficacy and tolerability; Phase I
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1-ADVATE+FRSW117(25 IU/kg) (Experimental): Subjects received two treatments: 25 IU/kg ADVATE in the first period, followed by 25 IU/kg FRSW117 in the second period, with a washout period before each treatment.
  Interventions: Drug: ADVATE; Drug: FRSW117
- Arm 2-ADVATE+FRSW117( 50 IU/kg) (Experimental): Subjects received two treatments: 50 IU/kg ADVATE in the first period, followed by 50 IU/kg FRSW117 in the second period, with a washout period before each treatment.
  Interventions: Drug: ADVATE; Drug: FRSW117

INTERVENTIONS:
Drug: ADVATE — a single dose.
Drug: FRSW117 — a single dose.
  Other Names: PEG Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection

SUMMARY:
The primary objectives of the study are to evaluate the Pharmacokinetics，Safety and tolerability of PEG Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection (FRSW117) in patients with severe hemophilia A.

The secondary objectives are to monitor anti-durg antibodies and anti-PEG antibodies levels in patients with severe hemophilia A

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically confirmed hemophilia A (coagulation factor VIII <1%) and previous medical records confirming exposure to coagulation factor VIII for ≥150 days (EDs ≥150).
* Non-immunodeficient, with some immunity (CD4 > 200/μL).
* Platelet count >100×10^9/L.
* Normal prothrombin time (PT) or international normalized ratio (INR) <1.3.
* Negative lupus anticoagulant.
* Fully understand, informed about this study and sign the informed consent form, voluntarily participate in the clinical study and have the ability to complete all study procedures

Exclusion Criteria:

* Hypersensitivity to the test substance or its excipients (including rodent or hamster protein).
* Pre-existing hypersensitivity or allergic reactions to FVIII or IgG2 injection therapy.
* Positive FVIII inhibitor at screening (≥0.6 BU/mL), or previous history of FVIII inhibitor Positive history, or family history of inhibitors.
* Patients with other coagulation disorders in addition to hemophilia A.
* The results of vWF antigen examination lower than normal.
* Severe anemia and need blood transfusion (hemoglobin < 60g/L).
* Patients who have received any standard half-lives FVIII formulations (e.g., Kogenate, Kovaltry, Advate, Xyntha, etc.) or received any other half-life-extending FVIII formulations within 4 days or 5 half-lives (whichever is longer) before administration.
* Patients who had used emecizumab within 6 months prior to administration.
* Patients with fever, upper respiratory tract infection or allergy symptoms within the previous 2 weeks before screening.
* Suffer from other diseases that may increase the risk of bleeding or the risk of thrombosis.
* Severe cardiovascular and cerebrovascular diseases: such as cerebral hemorrhage, stroke, myocardial infarction, unstable angina pectoris, congestive heart failure(the current New York Heart Association cardiac function grade III, Hypertension that cannot be controlled with drug treatment: systolic blood pressure> 160 mmHg or diastolic blood pressure> 95 mmHg.
* Clinically significant of other systematic diseases: alcoholism, drug abuse, mental disorders and mental retardation.
* Significant hepatic or renal impairment (ALT and AST > 2×ULN; serum bilirubin level > 3 × upper limit of normal (ULN)).
* Abnormal kidney function: BUN > 2×ULN, Cr > 2.0mg/dL.
* One or more clinically significant tests for Hepatitis B Virus Surface Antigen, Human Immunodeficiency Virus (HIV), Antisyphilitic spirulina (TPHA) and Hepatitis C Virus (HCV) Antibody.
* Patients who received any anticoagulant or antiplatelet therapy within a week prior screening or need to receive an anticoagulant or antiplatelet therapy during the period of clinical trials.
* Systemic immunomodulators (e.g., corticosteroids [equivalent dose of 10 mg/ day prednisone], A-interferon, immunoglobulin, cyclophosphamide, cyclosporine, etc.) were used within 14 days prior to administration or during the study period.
* Patients having major surgery or receiving blood or blood components transfusion within 4 weeks prior screening or having planned major surgery schedule during the study.
* Patients who previously participated in the other clinical trials within a month prior screening.
* Any life-threatening disease or condition which, according to the investigator's judgment, could not benefit from the trial participation.
* Patient who is considered by the other investigators not suitable for clinical study.

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2021-10-17 (Actual); Study Completion 2021-10-17 (Actual)

PRIMARY OUTCOMES:
Cmax from time 0 to the last data point for FRSW117 Measured by One-Stage Clotting Assay. | Pre-dose to 216 hours after the end of the infusion for Arm1; Pre-dose to 288 hours after the end of the infusion for Arm2
  Maximum plasma activity during a dosing interval for participants.
Arm1 - T½ from time 0 to the last data point for FRSW117 Measured by One-Stage Clotting Assay. | Pre-dose to 216 hours after the end of the infusion for Arm1; Pre-dose to 288 hours after the end of the infusion for Arm2
  Time required for the activity of the drug to reach half of its original value for participants.
Arm1 - CL from time 0 to the last data point for FRSW117 Measured by One-Stage Clotting Assay. | Pre-dose to 216 hours after the end of the infusion for Arm1; Pre-dose to 288 hours after the end of the infusion for Arm2
  Rate at which the body removes the drug, measured as the volume of the plasma cleared of drug per unit time per unit weight for participants.
Arm1 - MRT from time 0 to the last data point for FRSW117 Measured by One-Stage Clotting Assay. | Pre-dose to 216 hours after the end of the infusion for Arm1; Pre-dose to 288 hours after the end of the infusion for Arm2
  The average time that a drug molecule is present in the systemic circulation for participants.
Arm1 - Incremental recovery from time 0 to the last data point for FRSW117 Measured by One-Stage Clotting Assay. | Pre-dose to 216 hours after the end of the infusion forArm1; Pre-dose to 288 hours after the end of the infusion for Arm2
  The rise in FVIII activity in IU/dL per unit dose administered in IU/kg for participants.
Arm1 - Cmax from time 0 to the last data point for ADVATE Measured by One-Stage Clotting Assay. | Pre-dose to 72 hours after the end of the infusion for Arm1; Pre-dose to120 hours after the end of the infusion for Arm2
  Maximum plasma activity during a dosing interval for participants.
Arm1 - T½ from time 0 to the last data point for ADVATE Measured by One-Stage Clotting Assay. | Pre-dose to 72 hours after the end of the infusion for Arm1; Pre-dose to120 hours after the end of the infusion for Arm2
  Time required for the activity of the drug to reach half of its original value for participants.
Arm1 - CL from time 0 to the last data point for ADVATE Measured by One-Stage Clotting Assay. | Pre-dose to 72 hours after the end of the infusion for Arm1; Pre-dose to120 hours after the end of the infusion for Arm2
  Rate at which the body removes the drug, measured as the volume of the plasma cleared of drug per unit time per unit weight for participants.
Arm1 - MRT from time 0 to the last data point for ADVATE Measured by One-Stage Clotting Assay. | Pre-dose to 72 hours after the end of the infusion for Arm1; Pre-dose to120 hours after the end of the infusion for Arm2
  The average time that a drug molecule is present in the systemic circulation for participants.
Arm1 - Incremental recovery from time 0 to the last data point for ADVATE Measured by One-Stage Clotting Assay. | Pre-dose to 72 hours after the end of the infusion for Arm1; Pre-dose to120 hours after the end of the infusion for Arm2
  The rise in FVIII activity in IU/dL per unit dose administered in IU/kg for participants.
Number of participants with treatment-emergent adverse events (TEAEs). | assessed up to four weeks after FRSW117 administration.
  Adverse events in the study were classified and evaluated according to the National Cancer Institute's Common Terminology for Adverse Events (NCI CTCAE V5.0).

SECONDARY OUTCOMES:
Evaluation of the level of anti-PEG-rFⅧFc antibody production in participants | assessed up to four weeks after FRSW117 administration.
Evaluation of the level of anti-PEG antibody production in participants | assessed up to four weeks after FRSW117 administration.
Number of participants with inhibitor development. | assessed up to four weeks after FRSW117 administration.
  Number of participants who developed a positive FVIII inhibitor level (≥0.6 Bethesda unit [BU]) during the study was summarized and classified as participants developing low titer inhibitor (i.e. ≤ 5.0 BU) and participants developing high titer inhibitor (i.e. > 5.0 BU).

CONTACTS AND LOCATIONS:
Overall Officials: Renchi Yang, PhD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences & Peking Union Medical College.
Locations (4):
- China (4):
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangzhou
  - People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Jinan central hospital, Jinan, Shandong
  - Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences & Peking Union Medical College., Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No